CLINICAL TRIAL: NCT05197868
Title: Applied Forces During Neonatal Intubation: a Randomized Crossover Mannequin Study
Brief Title: Applied Forces During Neonatal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NEOUNIPD1
Record Dates: First submitted 2021-11-28; First posted 2022-01-20 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Intubation; Training; Neonate; Manikin
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intubation with traditional laryngoscope (Active Comparator): Participants will be required to intubate the manikin by using a traditional laryngoscope
  Interventions: Procedure: Intubation with traditional laryngoscope
- Intubation with a straight blade video laryngoscope (Experimental): Participants will be required to intubate the manikin by using a straight blade video laryngoscope
  Interventions: Procedure: Intubation with a straight blade video laryngoscope
- Intubation with hyper-angulated video laryngoscope (Experimental): Participants will be required to intubate the manikin by using a hyper-angulated video laryngoscope
  Interventions: Procedure: Intubation with a hyper-angulated video laryngoscope

INTERVENTIONS:
Procedure: Intubation with traditional laryngoscope — Participants will be invited to intubate the mannequin with a traditional laryngoscope
  Arms: Intubation with traditional laryngoscope
Procedure: Intubation with a straight blade video laryngoscope — Intubation with a straight blade video laryngoscope
  Arms: Intubation with a straight blade video laryngoscope
Procedure: Intubation with a hyper-angulated video laryngoscope — Participants will be asked to intubate the mannequin with a hyper-angulated video laryngoscope
  Arms: Intubation with hyper-angulated video laryngoscope

SUMMARY:
This study will be to compare the forces applied to mannequin airways (at epiglottis and at palate) during direct laryngoscopy and indirect video laryngoscopy with two kinds of blades (straight blade and hyper-angulated blade)

DETAILED DESCRIPTION:
This is a randomized controlled crossover trial of intubation with three laryngoscope devices in a neonatal manikin model. Level III NICU and PICU consultants, pediatric residents, anesthesiology consultants, and anesthesiology residents will be eligible to participate in the study. Participants in the ABC arm will be assigned to perform the intubation with a traditional laryngoscope (A), followed by the intubation with a straight blade video laryngoscope (B) and by the intubation with hyper-angulated video laryngoscope (C). Participants in different arms will be assigned to perform the intubations in different sequences (BCA/CAB/ACB/BAC/CBA). The primary outcome measure will be the forces applied to mannequin oro-tracheal tissues during intubation with the three kinds of tools. The secondary outcome measures will be the perceived workload during intubation and intubation time with the traditional laryngoscope and the video laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU and PICU consultants, pediatric residents, anesthesiology consultants, and anesthesiology residents will be eligible to participate in the study.

Exclusion Criteria:

* Refusal to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Forces applied to the epiglottis | 5 minutes
  The peak force (maximum force, expressed as Newton) applied on the epiglottis during intubation will be recorded by sensors positioned on the tip of the laryngoscope's blade.

SECONDARY OUTCOMES:
Forces applied to the palate | 5 minutes
  The peak force (maximum force, expressed as Newton) applied on the palate during intubation will be recorded by sensors positioned on the posterior side of the laryngoscope's blade.
Perceived workload during intubation | 20 minutes
  Participants will be asked to report their perceived workload during intubation by using a validated tool
Time of intubation | 5 minutes
  Time elapsed frmo insertion of the laryngoscope in the mouth to his removal

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balaban O, Tobias JD. Videolaryngoscopy in Neonates, Infants, and Children. Pediatr Crit Care Med. 2017 May;18(5):477-485. doi: 10.1097/PCC.0000000000001128. PMID 28319487
- [Result] Gordon JK, Bertram VE, Cavallin F, Parotto M, Cooper RM. Direct versus indirect laryngoscopy using a Macintosh video laryngoscope: a mannequin study comparing applied forces. Can J Anaesth. 2020 May;67(5):515-520. doi: 10.1007/s12630-020-01583-x. Epub 2020 Mar 9. PMID 32152886
- [Result] Pouppirt NR, Nassar R, Napolitano N, Nawab U, Nishisaki A, Nadkarni V, Ades A, Foglia EE. Association Between Video Laryngoscopy and Adverse Tracheal Intubation-Associated Events in the Neonatal Intensive Care Unit. J Pediatr. 2018 Oct;201:281-284.e1. doi: 10.1016/j.jpeds.2018.05.046. Epub 2018 Jul 3. PMID 29980290
- [Derived] Cavallin F, Sala C, Maglio S, Bua B, Villani PE, Menciassi A, Tognarelli S, Trevisanuto D. Applied forces with direct versus indirect laryngoscopy in neonatal intubation: a randomized crossover mannequin study. Can J Anaesth. 2023 May;70(5):861-868. doi: 10.1007/s12630-023-02402-9. Epub 2023 Feb 14. PMID 36788198